CLINICAL TRIAL: NCT02573987
Title: MEOPA (Equimolar Mix of Oxygen and Nitrogen Monoxide) Versus Local Anesthesia for Analgesia During Chorionic Villus Sampling.
Brief Title: MEOPA Versus Local Anesthesia for Analgesia During Chorionic Villus Sampling.
Acronym: MELIBIO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, Raoul Desbriere, Dr Desbriere, Hospital St. Joseph, Marseille, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A121414-31
Record Dates: First submitted 2015-09-17; First posted 2015-10-12 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Oxygen; Meopa; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen/nitrous oxide equimolar mix (Active Comparator): 96 participants undergoing chorionic villi sampling. self administered inhalation of equimolar mixture of oxygen and nitrous oxide (MEOPA)
  Interventions: Drug: Oxygen/nitrous oxide equimolar mix
- Lidocaine (Active Comparator): 96 participants undergoing chorionic villi sampling infiltrative local anaesthesia of 1% lidocaine
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Oxygen/nitrous oxide equimolar mix — an experimental strategy inhalation by means of a breathing mask diffusing MEOPA
  Other Names: MEOPA
  Arms: Oxygen/nitrous oxide equimolar mix
Drug: Lidocaine — standard strategy by local injection anesthesia of lidocaine
  Arms: Lidocaine

SUMMARY:
determine if efficiency of MEOPA anesthesia is at least equivalent to local anesthetics into the chorionic villus sampling in the first trimester of pregnancy

DETAILED DESCRIPTION:
Compare anxiety discomfort and side effects

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* 18 and over
* monofetal pregnancy
* chorionic villus sampling medical indication without contra indication
* informed consent signature

Exclusion Criteria:

* pregnant under 18
* multiple pregnancies
* pregnancy inferior 11 aw
* no informed consent signature

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-12-27 (Actual)

PRIMARY OUTCOMES:
Analgesia efficiency | 5 min after procedure
  assessment of pain with visual analog scale

SECONDARY OUTCOMES:
assessment of anxiety | 5 min after biopsy
  assessment of anxiety with visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Desbriere, MD, Principal Investigator — Hôpital st Joseph Marseille France
Locations (1):
- Hôpital St Joseph, Marseille, France